CLINICAL TRIAL: NCT00509652
Title: Therapeutic Effect of Erythrocyte Apheresis as Compared to Full Blood Phlebotomy in Patients With Hereditary Hemochromatosis
Brief Title: Erythrocyte Apheresis Versus Phlebotomy in Hemochromatosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Helse Fonna (Other); Haukeland University Hospital (Other); University Hospital, Akershus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSD13903
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Hemochromatosis
Keywords: Hemochromatosis; Primary hemochromatosis; Hereditary hemochromatosis; Therapy; Erythrocyte apheresis; Phlebotomy; Apheresis; Efficacy
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Erythrocyte apheresis
  Interventions: Procedure: Arm 1: Erythrocyte apheresis
- Arm 2 (Active Comparator): Phlebotomy
  Interventions: Procedure: Arm 2: Whole blood phlebotomy

INTERVENTIONS:
Procedure: Arm 1: Erythrocyte apheresis — Erythrocyte apheresis
  Arms: Arm 1
Procedure: Arm 2: Whole blood phlebotomy — Traditional whole blood phlebotomy
  Arms: Arm 2

SUMMARY:
Primary hemochromatosis is the most frequent hereditary condition in Scandinavia. The condition may result in serious organ damage which can be prevented by therapy, but only few patients develop such organ damage. The optimal treatment, therefore, is still a matter of discussion Prevention of organ damage has traditionally been accomplished by drawing of full blood (phlebotomy), which has to be frequently repeated during the initial phase and then continued indefinitely as a maintenance treatment. The removed amount of iron may be increased two- or threefold for each procedure by using modern equipment for selective removal of red blood cells (red cell apheresis). Possible drawbacks of this technique may be higher costs, prolonged time for each therapeutic procedure, and certain requirements to the patients. The possible advantages are the reduced number of therapeutic procedures and less strain for the patient. No larger, randomized study has been published in order to determine which method should be preferred.

This study is a controlled trial in which participating patients are asked to be randomized to red cell apheresis or traditional phlebotomy. Each group will be followed by means of well-defined assessments in order to explore possible advantages and disadvantages of each method in order to establish what type of treatment should be recommended.

DETAILED DESCRIPTION:
Introduction Primary hemochromatosis is the most frequent hereditary condition in Scandinavia. The condition may result in serious organ damage which can be prevented by therapy, but only few patients develop such organ damage. Provided the lack of more exact knowledge of which patients should be treated, we have based our inclusion criteria on the guidelines published by the Norwegian Society of Hematology. However, the criteria for ferritin levels have been set at 300 micrograms/L for patients who are homozygous for the C282Y mutation, and also heterozygous individuals will be included if ferritin is higher than 500 micrograms/L.

Furthermore, the optimal treatment method is still a matter of discussion. Prevention of organ damage has traditionally been accomplished by whole blood phlebotomy, which has to be frequently repeated during the initial phase and then continued indefinitely as a maintenance treatment. The removed amount of iron may be increased two- or threefold for each procedure by using modern equipment for selective withdrawal of red blood cells (erythrocyte apheresis). Possible drawbacks of this technique may be higher costs, prolonged time for each therapeutic procedure, and certain requirements to the patients. The possible advantages are the reduced number of therapeutic procedures and less strain for the patient. No larger, randomized study has been published in order to determine which method should be preferred.

Hypothesis: A more rapid decline of primary endpoints (see below) can be achieved by erythrocyte apheresis as compared to traditional phlebotomy, without significant disadvantages.

Design The trial is prospective, randomized and open. Eligible patients are randomized to erythrocyte apheresis and phlebotomy.

Endpoints Primary endpoints Decline of ferritin levels and transferrin saturation.

Secondary endpoints and other variables to be studied Decline in hemoglobin levels. Discomfort during the therapeutic procedure. Any changes in EVF, blood cell counts or albumin and CRP levels. Certain well-defined financial costs: consumed material, technician working time.

Inclusion criteria

1. Diagnosis

   1. Individuals who art homozygous for C282Y or H63D or "compound heterozygous" for these tow variants and have ferritin levels higher than 300 micrograms/L or transferrin saturation higher than 50%.
   2. Individuals heterozygous for C282Y or H63D if ferritin levels higher than 500 micrograms/L or transferrin saturation higher than 50%.
2. Requirements to the patient Body weight higher than 65 kg and initial hemoglobin level higher than 12 g/dL.

Treatment schedule Following randomization to either apheresis or phlebotomy, patients are treated until ferritin levels have declined to below 50 micrograms/L and they are then followed for one year. Patients randomized to apheresis are treated every second week, whereas patients in the phlebotomy group are treated weekly. Prolongation of the interval is permitted in both groups in case of well-defined clinical indications. Any prolongation is to be recorded along with the clinical indication.

Follow-up Clinical symptoms, body weight, laboratory findings (Hemoglobin levels; blood cell counts; levels of iron, transferrin, ferritin, albumin and IgG; serologic assessments for hepatitis viruses, CMV and HIV), discomfort during the therapeutic procedure, duration of each procedure, costs for consumed material, working time of the technician for each procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis

   * Individuals who art homozygous for C282Y or H63D or "compound heterozygous" for these tow variants and have ferritin levels higher than 300 micrograms/L or transferrin saturation higher than 50%.
   * Individuals heterozygous for C282Y or H63D if ferritin levels higher than 500 micrograms/L or transferrin saturation higher than 50%.
2. Requirements to the patient Body weight higher than 65 kg and initial hemoglobin level higher than 12 g/dL.

Exclusion Criteria:

1. Contra-indications to either treatment modality
2. Patients who are not able to co-operate
3. Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2006-01; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Decline in ferritin levels and transferrin saturation

SECONDARY OUTCOMES:
Decline in hemoglobin levels
Patient discomfort during therapeutic procedure
Time consumption
Costs

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Sundic, MD, Principal Investigator — Department of Immunology and Transfusion Medicine, Haugesund Hospital; Sigbjorn Berentsen, MD, PhD, Study Chair — Department of Medicine, Haugesund Hospital; Tor Hervig, MD, PhD, Study Chair — Department of Transfusion Medicine, Haukeland University Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Department of Transfusion Medicine, Bergen
  - Haugesund Hospital, Department of Immunology and Transfusion Medicine, Haugesund
  - Akershus University Hospital (AHUS), Department of Transfusion Medicine, Nordbyhagen

REFERENCES:
- [Background] Asberg A, Hveem K, Thorstensen K, Ellekjter E, Kannelonning K, Fjosne U, Halvorsen TB, Smethurst HB, Sagen E, Bjerve KS. Screening for hemochromatosis: high prevalence and low morbidity in an unselected population of 65,238 persons. Scand J Gastroenterol. 2001 Oct;36(10):1108-15. doi: 10.1080/003655201750422747. PMID 11589387
- [Background] Muncunill J, Vaquer P, Galmes A, Obrador A, Parera M, Bargay J, Besalduch J. In hereditary hemochromatosis, red cell apheresis removes excess iron twice as fast as manual whole blood phlebotomy. J Clin Apher. 2002;17(2):88-92. doi: 10.1002/jca.10024. PMID 12210712
- [Background] Rombout-Sestrienkova E, van Noord PA, van Deursen CT, Sybesma BJ, Nillesen-Meertens AE, Koek GH. Therapeutic erythrocytapheresis versus phlebotomy in the initial treatment of hereditary hemochromatosis - A pilot study. Transfus Apher Sci. 2007 Jun;36(3):261-7. doi: 10.1016/j.transci.2007.03.005. Epub 2007 Jun 13. PMID 17569592
- [Background] Knutsen, H. & Hammerstrom, J. Handlingsprogram for hemokromatose [Norwegian national program for treatment of haemochromatosis]. http://www.legeforeningen.no/asset/22333/1/22333_1.doc . 2003. Norwegian Society of Haematology.
- [Background] Telset BIV. Behandling av hereditær hemokromatose: fullblodstapping eller erytrocyttaferese? [Treatment of hereditary haemochromatosis: whole blood phlebotomy or red cell apheresis?] Master Thesis. Bergen: Faculty of Medicine, University of Bergen, 2004